CLINICAL TRIAL: NCT06853860
Title: Comparison of the Effects of Reflexology and Classical Hand Massage on Pain, Anxiety, and Vital Signs in Patients After Coronary Angiography
Brief Title: Effects of Hand Massage Applied With Two Different Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Necibe Dağcan, Assistant Professor of Nursing, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KutahyaHSU-NECİBE-DAĞCAN-0006
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-08

CONDITIONS: Angiopathy, Peripheral; Pain, Acute; Reflexology
MeSH Terms: conditions — Peripheral Vascular Diseases; Acute Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: This study is a double-blind randomized controlled trial planned to investigate the effects of hand massage applied with two different methods on pain, anxiety and physiological parameters in patients undergoing coronary angiography.
Who Masked: Outcomes Assessor
Masking Description: Patients will be divided into experimental and control groups. Patients will know that they are participating in the study and the interventions that will be applied to them, but they will be blinded by not knowing which group they are in. The study data will be collected by a second researcher who is blinded to the groups. In the statistical analysis of the data, the groups will be labeled as group 1 and group 2, and the third researcher will be blinded when evaluating the results. Thus, the third researcher will be blinded to the study groups. In order to avoid bias in the evaluation of the results, the first researcher who is not blinded will not participate in any stage of the evaluation process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- reflexology group (Experimental): reflexology group
  Interventions: Other: reflexology massage
- Classic hand massage group (Placebo Comparator): Classic hand massage group
  Interventions: Other: classic hand massage

INTERVENTIONS:
Other: reflexology massage — classic hand massage
  Arms: reflexology group
Other: classic hand massage — classic hand massage
  Arms: Classic hand massage group

SUMMARY:
There is no study finding examining the effects of the classical hand massage and hand reflexology massage methods on pain, anxiety and physiological parameters after coronary angiography. Therefore, the aim of this study is to examine the effects of reflexology hand massage and classical hand massage on pain, anxiety and physiological parameters after coronary angiography.

DETAILED DESCRIPTION:
There is no study finding examining the effects of the classical hand massage and hand reflexology massage methods on pain, anxiety and physiological parameters after coronary angiography.

ELIGIBILITY:
Inclusion Criteria:

* • Patients who are over 18 years old

  * Can speak Turkish
  * Agree to participate in the study
  * Have not undergone emergency coronary angiography
  * Have not consumed coffee or hypnotic drugs at least 12 hours before
  * Have no history of chronic pain (e.g. arthritis)
  * Are not addicted to alcohol or drugs
  * Have no psychological problems (such as depression, anxiety disorder)
  * Have no problem with having their hands massaged; those who do not have any skin lesions, sensory and motor disorders, amputations, burns, or pathological diseases related to muscles and bones
  * Have not used anxiolytics

Exclusion Criteria:

* • Those who do not volunteer to participate in the study

  * Those who have any skin lesions, burns, open wounds, muscle and bone pathological diseases on their hands,
  * Those who develop delirium during the follow-up period
  * Those who develop complications after coronary angiography (such as bleeding, etc.)
  * Arrhythmia
  * Hemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Average Pain Score on Visual Analog Scale (VAS) | 0 hour (baseline), 1st hour, 2nd hour, 3rd hour
  Pain will be measured using the Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (severe pain). Higher scores indicate more severe pain.
State Anxiety Scale Mean Score | 0 hour (baseline), 1st hour, 2nd hour, 3rd hour
  Anxiety will be measured using the State Anxiety Scale, a validated questionnaire assessing current anxiety levels. Higher scores indicate higher levels of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu NAL, PhD, Study Director — Kütahya Health Sciences University, Faculty of Health Sciences; Mehmet Ali ASTARCIOĞLU, Prof., Study Director — Kütahya Health Sciences University, Faculty of Health Sciences
Locations (1):
- Necibe, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No